CLINICAL TRIAL: NCT06688123
Title: A Randomized, Open-label, Treat-to-target, Parallel-controlled, Phase II Clinical Study to Evaluate the Efficacy and Safety of SHR-3167 and Insulin Glargine in Patients With Type 2 Diabetes Mellitus With Metformin Alone or in Combination With SGLT2 Inhibitors
Brief Title: Efficacy and Safety of SHR-3167 and Insulin Glargine in Type 2 Diabetes Subjects
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3167-201
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-3167 group A (Experimental)
  Interventions: Drug: SHR-3167
- SHR-3167 group B (Experimental)
  Interventions: Drug: SHR-3167
- Insulin glargine group (Active Comparator)
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: SHR-3167 — Dose level 1.
  Arms: SHR-3167 group A
Drug: SHR-3167 — Dose level 2.
  Arms: SHR-3167 group B
Drug: Insulin glargine — Dose level 3.
  Arms: Insulin glargine group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SHR-3167 compared with insulin glargine after treatment in insulin naïve subjects with type 2 diabetes treated with metformin alone or in combination with SGLT2 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Diagnosed with type 2 diabetes mellitus ≥ 6 months prior to the day of screening.
3. A stable dose of metformin alone or in combination with a stable dose of a SGLT2 inhibitor for 3 months prior to screening.
4. Body mass index (BMI): 18.5~35.0 kg/m2.
5. HbA1c of 7.5%~10.0% as assessed by the local laboratory.
6. Insulin naïve.
7. Female subjects and partners of male subjects who are of childbearing potential, have no fertility plan and agree to take highly effective contraceptive measures within 6 months after signing the informed consent form to the last dose, and have no plans to donate eggs/sperm; Female subjects of childbearing potential have a negative pregnancy test during the screening period and are not lactating.

Exclusion Criteria:

1. Electrocardiogram (ECG) results show clinically significant abnormalities that may affect the safety of the subject.
2. Poor blood pressure control at screening.
3. Diagnosis or suspicion of type 1 diabetes mellitus, latent autoimmune diabetes mellitus in adult (LADA)，other special types of diabetes or secondary diabetes mellitus.
4. ≥1 episode of severe hypoglycemia or asymptomatic hypoglycemia within 6 months prior to screening, or recurrent hypoglycemic events within 1 month prior to screening.
5. History of diabetic ketoacidosis or hyperosmolar hyperglycemic state due to hyperglycemia within 6 months prior to screening.
6. Presence of acute or chronic hepatitis, cirrhosis, or other serious liver disease other than non-alcoholic fatty liver disease.
7. Those who have a history of severe cardiovascular and cerebrovascular diseases within 6 months before screening.
8. Malignancy or history of malignancy within 5 years prior to screening.
9. Received any diabetes mellitus or weight-loss medication outside the inclusion criteria within 3 months prior to screening.
10. Participation in a clinical trial of any drug or medical device within 3 months prior to screening.
11. Any other condition judged by the investigator to be likely to affect the subject's safety or interfere with the evaluation of trial results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to week 20 in HbA1c (HemoglobinA1c) | Week 0 to week 20.
  Change from baseline in HbA1c after 20 weeks of treatment.

SECONDARY OUTCOMES:
Percentage of participants achieving HbA1c<7.0% | Week 0 to week 20.
Change from baseline to week 20 in fasting plasma glucose (FPG) | Week 0 to week 20.
Change from baseline to week 20 in self-measured blood glucose (SMBG) before breakfast | Week 0 to week 20.
Number of adverse events (AEs) during the trial | Week 0 to week 24.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided